CLINICAL TRIAL: NCT02291822
Title: The Safety and Efficacy of MULTIHANCE at the Dose of 0.10 mmol/kg in Magnetic Resonance Imaging of the Central Nervous System in Pediatric Patients Who Are Less Than 2 Years of Age
Brief Title: Retrospective Study of MRI in Pediatric Patients
Status: Completed | Type: Observational
Sponsor: Bracco Diagnostics, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: MH-150
Record Dates: First submitted 2014-11-06; First posted 2014-11-17 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2015-05

CONDITIONS: Central Nervous System Disease; Central Nervous System Neoplasms
MeSH Terms: conditions — Central Nervous System Diseases; Central Nervous System Neoplasms | interventions — gadobenic acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gadobenate Dimeglumine — gadolinium contrast agent
  Other Names: MultiHance

SUMMARY:
Collection of already existing data and images for patients < 2 years of age having MultiHance administration for a MRI of the brain or spine. MR Images will be reviewed during a prospectively designed blinded reading of the images.

ELIGIBILITY:
Inclusion Criteria:

* Male or female less than 2 years of age at the time of the MRI with MultiHance injection at a dose of 0.1 mmol/kg (± 25% in volume administered)
* Has available demographic and safety data
* Has documented known or highly suspected enhancing disease of the CNS (brain/spine) and previously underwent a cranial or spinal MR examination requiring an injection of MULTIHANCE contrast agent
* Has both pre and post dose T1 SE/FSE and/or GRE and T2 SE/FSE, and FLAIR MR images (when available) for submission to sponsor or designee to be evaluated in a fully blinded read
* Has a documented dose of MultiHance administered for their MRI exam and/or volume (mL) and weight of the patient available to be used to calculate the dose of MultiHance that was administered

Exclusion Criteria:

* Any patient who does not fulfill all of the inclusion criteria

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients less than 2 years of age who have previously undergone a MRI of the brain or spine with MultiHance
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Border delineation of lesions | Immediately post dose - Day 1
  Unenhanced MRI and contrast enhanced MRI are superior to unenhanced MRI alone in terms of lesion border delineation
Visualization of internal morphology of lesions | Immediately post dose - Day 1
  Unenhanced MRI and contrast enhanced MRI are superior to unenhanced MRI alone in terms of visualization of internal morphology of the lesion(s)
Contrast enhancement of lesions | Immediately post dose- Day 1
  Unenhanced MRI and contrast enhanced MRI are superior to unenhanced MRI alone in terms of contrast enhancement of lesions

CONTACTS AND LOCATIONS:
Overall Officials: Gianpaolo Priovano, M.D., Study Director — Bracco Diagnostics, Inc